CLINICAL TRIAL: NCT03571360
Title: Expression/DNA Methylation of Cancer Testis Antigens May Predict Response to Pembrolizumab in Non-small Cell Lung Cancer Patients
Brief Title: CTA Expression/Methylation and Response to Pembrolizumab of NSCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerwin Heller, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-000689-30
Record Dates: First submitted 2018-06-12; First posted 2018-06-27 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Other): Pembrolizumab 200 mg i.v., every 3 weeks, maximum of 2 years
  Interventions: Other: PD-L1 positive vs PD-L1 negative NSCLC patients

INTERVENTIONS:
Other: PD-L1 positive vs PD-L1 negative NSCLC patients — Genomic analyses of PD-L1 positive vs PD-L1 negative NSCLC patients

SUMMARY:
Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. KeytrudaTM (pembrolizumab) has been approved by the FDA and the EMA for the therapy of with chemotherapy pretreated NSCLC patients with PD-L1 expression (TPS ≥ 1%) on tumor cells. In addition, pembrolizumab was approved for the first line treatment of metastatic NSCLC patients with high PD-L1 expression (TPS ≥ 50%) on tumor cells. Pembrolizumab will be given in a flat dose of 200 mg i.v. every 3 weeks until disease progression, toxicity or patient withdrawal for a maximum of 2 years. Patients with untreated advanced stage lung adenocarcinoma, without an EGFR mutation or ALK translocation, will be included.

ELIGIBILITY:
Subject inclusion criteria:

1. Have an untreated lung adenocarcinoma of advanced stage.
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be at least 18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1.
6. Have a performance status of ≤1 on the ECOG Performance Scale
7. Demonstrate adequate organ function
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Subject exclusion criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has received radiotherapy within 14 days before the first dose of study treatment or received lung radiation therapy of > 30 Gy within 6 months before the first dose of study treatment.
3. Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
4. Has had an allogeneic tissue/solid organ transplant.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has a known history of active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has had prior chemotherapy, targeted small molecule therapy or therapy with an anticancer monoclonal antibody.
9. Has had radiation therapy within 2 weeks prior to study Day 1.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or CTLA-4 agent.
19. Has a known history of Human Immunodeficiency Virus (HIV).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C.
21. Has received a live vaccine within 30 days of planned start of study therapy.
22. Evidence of interstitial lung disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-01-14 (Estimated); Study Completion 2021-07-14 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 months after start of treatment
  Complete and partial remission, stable disease; measured by computertomography; RECIST 1.1 criteria
PFS | Time from start of treatment to radiologically confirmed progressive disease or death due to any cause, whichever came first, assessed up to 24 months.
  Distribution of PFS of patients

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Zöchbauer-Müller, MD, Principal Investigator — Medical University of Vienna, Vienna, Austria
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No